CLINICAL TRIAL: NCT00719628
Title: Depth of Anaesthesia and Presence of Postoperative Cognitive Dysfunction
Brief Title: Depth of Anaesthesia and Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Jacob Steinmetz, Dep Anaesthesia, HOC 4231, Rigshospitalet
Other Study IDs: JAS-001
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Cognitive Dysfunction
Keywords: Postoperative; Cognitive; Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate if there is an association between the depth of anaesthesia and the presence of cognitive deterioration after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60
* Surgery in general anesthesia
* surgery > 1 hour
* ASA: 1-3

Exclusion Criteria:

* Dementia
* Excessive Use of alcohol or anxiolytics
* Unable to understand danish
* MMSE score < 24

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 60 years eligible for surgery
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
mean Cerebral state index in relation to postoperative cognitive dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Lars S Rasmussen, MD, PhD, Study Director — Dep anaesthesia, HOC, Rigshospitalet
Locations (1):
- Dep Anaesthesia, HOC, Rigshospitalet, Copenhagen, Denmark